CLINICAL TRIAL: NCT05376098
Title: A Temporal Study of Brain Motor Regions of Acute Ischemic Stroke Based on fNIRS
Brief Title: An fNIRS Study of Motor Cortical Activation in Stoke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: haojunwei7
Record Dates: First submitted 2022-04-01; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Motor rehabilitation; Brain regions; fNIRS
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators evaluate the activation and connectivity of patients' motor regions in the acute phase of ischemic stroke by fNIRS.

DETAILED DESCRIPTION:
This study aims to analyze the progress of brain recovery from upper-limb deficit due to acute ischemic stroke, using Functional Near-infrared Spectroscopy(fNIRS) as the main neural imaging method. Fifty patients having experienced a stroke onset within seven days will be recruited from the emergency room. The fNIRS signals will be recorded bilaterally over the contralateral sensorimotor cortex, the premotor area, the supplementary motor area, the primary motor cortex for 14 days after being diagnosed. Then compute activation and connectivity of the regions. The motor function data measured by the assessment scales, as well as the behavioral record during the fNIRS motor tasks will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ischemic stroke should meet the diagnostic criteria of the "China Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018".
* 18 years old≤ age ≤ 75 years old.
* Cerebral ischemic stroke onset within 7 days.
* First onset.
* Upper limb motor dysfunction.

Exclusion Criteria:

* Unstable vital signs.
* Complicated with other diseases in the nervous system.
* Combined with other serious disease states: circulatory system, respiratory system,
* motor system diseases, such as atrial fibrillation, heart failure, lung infection, severe liver and kidney dysfunction, lower limb venous thrombosis, etc.
* Upper limb dysfunction caused by other reasons, such as fractures, upper limb deformities, etc.
* Contraindicated to imaging tests, such as metal implantation, claustrophobia, and severe obesity.
* Those who cannot complete the examination due to other reasons, such as mental disorders, cognitive dysfunction, etc.
* Other causes: alcoholism; pregnancy; skull defects; soft tissue injuries at the site of examination; visual impairment, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke with upper limb motor dysfunction diagnosed and treated by the Xuanwu Hospital Capital Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
fNIRS characteristics of upper limb movement | 0-14 day
  The changes in brain oxygen levels are collected in two wavelengths, including 845 and 763 nanometers using a 44 channeled fNIRS machine. The data is used to determine the position of the activated area of the brain and functional connectivity during the movement. The locations of fNIRS channels on the skull of individuals are determined due to the observations on the cortical regions of interest (ROIs), namely the contralateral sensorimotor cortex (SMC), the contralateral premotor cortex (PMC) and primary motor cortex (M1), etc.
Assessment of upper limb function | 0-14 day
  Recording the quality and frequency of fNIRS motion tasks including grip and reach-out movements.
Assessment of upper limb function | 0-14 day
  Evaluating the motor function by Action Research Arm Test.
Assessment of upper limb function | 0-14 day
  Evaluating the motor function by Fugl-meyer assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China